CLINICAL TRIAL: NCT05794113
Title: Comparing the Use of a Mobile App for Surveillance of Adverse Events Following Influenza Immunization to a Web-Based Platform: a Randomized Controlled Trial
Brief Title: Comparing the Use of a Mobile App for Surveillance of Adverse Events Following Influenza Immunization to a Web-Based Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Ottawa Hospital (Other)
Responsible Party: Principal Investigator, Kumanan Wilson, Senior Scientist, The Ottawa Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: #20200591-01H
Record Dates: First submitted 2023-03-09; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Mobile Apps; Immunization; Adverse Event Following Immunisation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based notification arm (Active Comparator): All participants randomized to the web-based notification arm received the following web-based CANVAS notifications [4,5]. Briefly, participants received an email notifying them of their registration in the study. Eight days following their influenza vaccine, participants received an email with the survey link asking them to complete their online influenza vaccine safety survey. Participants received a reminder email on day 11 if they did not complete their survey.
  Interventions: Device: Web based notification
- Mobile app arm (Experimental): Participants randomized to the mobile app arm, received an email asking them to download the app and activate their account. Users who did not activate their account after 48 hours received a reminder email. Participants who activated their accounts, could spontaneously report an adverse event through the app, and were also notified of the day 8 survey through the app.
  Interventions: Device: Mobile app - CanImmunize

INTERVENTIONS:
Device: Mobile app - CanImmunize — Using a mobile app
  Arms: Mobile app arm
Device: Web based notification — Using a web-based version of a survey
  Arms: Web-based notification arm

SUMMARY:
Methods Study Procedures A two-centred randomized control trial (RCT) was conducted to evaluate the use of safety reporting via a mobile app compared to safety reporting via web-based CANVAS notifications amongst individuals receiving the influenza vaccine from October 6 to November 29, 2020 during the seasonal influenza vaccine campaign in Ottawa and Vancouver, Canada.

Individuals were recruited at the time of receiving their influenza vaccine. Eligibility criteria included the ability to speak English or French, having an active email address and telephone number, and being immunized with the seasonal influenza vaccine.

Randomization After study enrollment, participants were randomized to receive the online safety survey either through the mobile app or emailed a link to the online survey using a four-block randomization design.

Web-based notification arm All participants randomized to the web-based notification arm received the following web-based CANVAS notifications. Briefly, participants received an email notifying them of their registration in the study. Eight days following their influenza vaccine, participants received an email with the survey link asking them to complete their online influenza vaccine safety survey. Participants received a reminder email on day 11 if they did not complete their survey. Further details on CANVAS surveillance and description of the questionnaire can be found here.

Mobile app arm Participants randomized to the mobile app arm, received an email asking them to download the app and activate their account. Users who did not activate their account after 48 hours received a reminder email. Participants who activated their accounts, could spontaneously report an adverse event through the app, and were also notified of the day 8 survey through the app.

Eight days following their vaccination mobile app participants who activated their account received a push notification on their phone to complete their survey. A reminder push notice was sent out on day 11 to participants that had not yet competed the day 8 survey. On November 16, 2020 (mid-way through the recruitment period), additional email reminders in the mobile app arm were implemented on days 2, 4 and 6 to remind participants to register for the app. All participants received a day 8 email directing them to use their CANImmunize account to complete their influenza vaccine survey. Access to the survey link also was available in the email reminder.

ELIGIBILITY:
Inclusion Criteria:

* Speak English or French,
* Have an active email address and telephone • Immunized with the seasonal influenza vaccine
* Parents of children are eligible to participate after the first or second dose of vaccine

Exclusion Criteria:

* Those who do not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2408 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Useability | through study completion - average of 4 months
  Following completion of the safety survey, all participants were sent a separate link by email to complete a user experience survey. Participants were asked about their history of participating in the flu vaccine safety survey and whether they previously used the CANImmunize app. Using a Likert scale, participants were asked questions on (i) perceived ease of use, (ii) perceived usefulness, (iii) their attitudes and intention of use towards the platform and (iv) questions pertaining to vaccine confidence and safety.

CONTACTS AND LOCATIONS:
Overall Officials: Anne McCarthy, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bota AB, Bettinger JA, Sarfo-Mensah S, Lopez J, Smith DP, Atkinson KM, Bell C, Marty K, Serhan M, Zhu DT, McCarthy AE, Wilson K. Comparing the Use of a Mobile App and a Web-Based Notification Platform for Surveillance of Adverse Events Following Influenza Immunization: Randomized Controlled Trial. JMIR Public Health Surveill. 2023 May 8;9:e39700. doi: 10.2196/39700. PMID 37155240